

| Clinical Trial Protocol | |
|---|---|
| Protocol Title | Testing of Identification Markers for strokE |
| Acronym | TIME |
| NCT Identification | Not yet assigned |
| Number | |
| Version | 2.0 |
| Version date | 21st January 2020 |
| Study Sponsor | POCKiT diagnostics Ltd, Future Business Centre, CB4 2HY |
| | Cambridge, United Kingdom |
| Sponsor's Head of | Edoardo Gaude, PhD, POCKiT diagnostics Ltd |
| Clinical | |

# The University of Mississippi Medical Center 2500 North State Street Jackson, Mississippi 39216-4505

# **CONSENT FOR STORAGE AND FUTURE USE OF SAMPLES**

**Study Title**: Testing of Identification Markers for stroke (TIME)

**Sponsor**: POCKiT Diagnostics

Principal Investigator: Shashank Shekhar MD

Performance Site: University of Mississippi Medical Center

### **Introduction**

You are being invited to be in this observational research study because you were admitted to the Emergency Department with a suspected diagnosis of stroke. Please ask us about anything in this document or that we tell you that you do not understand.

### **Purpose**

We are doing this study to find new ways to diagnose stroke outside the hospital. This could be done by measuring certain blood molecules in patients right after they had a stroke. Early diagnosis is important in helping physicians provide the best possible treatment options. We will collect blood samples from patients with a suspected stroke. We will then measure the levels of certain blood molecules to understand if these can show the difference between people who had different types of stroke.

## **Procedures**

If you agree to participate in this study, you will provide a teaspoon of blood in addition to the blood drawn by the Emergency Department.

We would like to keep and store left over samples of your blood to use in future research studies. The samples may be used for commercial purposes.

We may use the samples to help us:

- Learn more about your disease.
- Learn more about other diseases or conditions.
- Find new ways to help people feel better.
- Learn how to treat, cure, or prevent the occurrence of stroke.

# <u>Risks</u>

There is very minimal risk to patients who participate. The risks of getting blood drawn include pain, bruising, or minor infection.

# **Benefits**

You will not receive a direct benefit from being in this research study. We hope to learn information that may help others in the future.

## **Compensation**

You will not be paid for participating in this study.

# **Voluntary Participation**

Your participation is voluntary. If you decide not to participate in this study you will not suffer a penalty or loss of benefits to which you are otherwise entitled.

## **Withdrawal**

You may choose to stop your participation in this study at any time. If you decide to withdraw the information already collected about you may still be used in this study but additional information will not be collected. Your decision to stop your participation will have no effect on the quality of medical care you receive at the University of Mississippi Medical Center.

## **Confidentiality**

Every effort will be made to keep the information we learn about you private. Study personnel, the Food and Drug Administration (FDA), the Office for Human Research Protections and University of Mississippi Medical Center's Institutional Review Board (IRB) and Office of Integrity and Compliance may review the study records. Any information which accompanies the sample when it leaves the hospital will have your name, address, and any other possible identifiable information removed so that you cannot be recognized from it.

#### **Protected Health Information**

Protected health information is any personal health information through which you can be identified. The information collected in this study includes: your final diagnosis, demographics, clinical data, and stroke scaling scores. By signing this consent document, you authorize Dr. Shekhar and his study staff to collect this information and use your records as necessary for this study.

#### **Number of Participants**

We expect 1,000 participants to enroll in this study here and 2,000 nationwide and internationally.

### Questions

If you have any questions about this study, please call Dr. Shekhar at 601-984-5500.

You will be given a copy of this consent document for your records if you agree to participate in this study.

# **Statement of Participation**

Your samples and some information about you will be stored in the UMMC Biobank and POCKiT Diagnostics. The samples and information may be used by other researchers, but no identifiers will be shared and no effort will be made to reconnect or re-identify your samples.

| no identifiers will be shared and no effort will be samples. | pe made to reconnect or re-identify your |
|---|---|
| It is your choice. You do not have to let us do not let us keep the left over samples. This par the study no matter what you decide. | |
| You may take, store and use samples related to my condition. | of my blood for future research studies |
| You may take, store and use samples studies do not have to be related to my condit | of my blood for future research studies. The ion. |
| I have been told about this study and the poss<br>voluntary and I may withdraw at any time with<br>am entitled, including medical care at the Univ | out any penalty or loss of benefits to which I |
| By signing this form I am not giving up any leg | gal rights I may have. |
| Printed name of Participant | _ |
| Signature of Participant | <br>Date |
| Printed name of person obtaining consent | |
| Signature of person obtaining consent | |
| <u>Date</u> | |

| I acknowledge that the participant identified above has been entered into this study, we properly obtained informed consent. |
|---|
| Signature of Principal Investigator |
| Date |